CLINICAL TRIAL: NCT04555044
Title: A Randomized, Double-Blind, Controlled, Clinical Trial to Evaluate the Risk of Developing Essential Fatty Acid Deficiency in Pediatric Patients, Including Neonates, Receiving Either Clinolipid (Lipid Injectable Emulsion, USP) 20% or Standard-of-Care Soybean Oil-Based Lipid Emulsion (Part A)
Brief Title: Pediatric Study to Evaluate Risk of Developing Essential Fatty Acid Deficiency When Receiving Clinolipid or Standard-of-Care Lipid Emulsion (Part A)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6344-001A
Record Dates: First submitted 2020-09-08; First posted 2020-09-18 (Actual); Results first posted 2023-12-27 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Essential Fatty Acid Deficiency (EFAD)
Keywords: Essential Fatty Acids (EFA); Parenteral Nutrition; Clinolipid/Clinoleic; Parenteral Nutrition Associated Cholestasis (PNAC); Parenteral Nutrition Associated Liver Disease (PNALD); Intestinal Failure Associated Liver Disease (IFALD); Phytosterols; Intralipid; Infants/Preterm Infants; FADS1 and FADS2; Short Bowel Syndrome; Cancer Nutrition; Olive Oil Emulsion; Soybean Oil Emulsion
MeSH Terms: conditions — Hyperphagia; Pena Shokeir syndrome, type 1; Short Bowel Syndrome | interventions — soybean oil, phospholipid emulsion

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Clinolipid (Experimental): Dosing based on American Academy of Pediatrics (AAP), American Academy Society for Parenteral and Enteral Nutrition (ASPEN), European Society for Paediatric Gastroenterology Hepatology and Nutrition (ESPGHAN)/ European Society for Parenteral and Enteral Nutrition (ESPEN)/ European Society of Paediatric Research (ESPR)/ Chinese Society for Parenteral and Enteral Nutrition (CSPEN) guidelines. Study treatment will be administered intravenously in the hospital setting from 7 up to 90 days using either a syringe pump or an infusion pump as appropriate for the daily volume of infusate. The flow rate will be prescribed by the Investigator to provide the daily dosage over 20 to 24 hours.
  Interventions: Drug: Clinolipid
- Intralipid (Active Comparator): Dosing based on AAP, ASPEN, ESPGHAN/ESPEN/ESPR/CSPEN guidelines. Study treatment will be administered intravenously in the hospital setting from 7 up to 90 days using either a syringe pump or an infusion pump as appropriate for the daily volume of infusate. The flow rate will be prescribed by the Investigator to provide the daily dosage over 20 to 24 hours.
  Interventions: Drug: Intralipid

INTERVENTIONS:
Drug: Clinolipid — Lipid injectable emulsion, USP 20%
  Arms: Clinolipid
Drug: Intralipid — Standard-of-Care Soybean Oil-Based Lipid Emulsion. 20% (lipid injectable emulsion, USP)
  Arms: Intralipid

SUMMARY:
This will be a descriptive study designed to evaluate the propensity for hospitalized pediatric patients treated adequately with Clinolipid or standard of care (Intralipid) from 7 up to 90 days to develop Essential Fatty Acid Deficiency (EFAD). Additionally, this study design will evaluate the safety and efficacy of using Clinolipid or Intralipid in a pediatric population.

ELIGIBILITY:
Inclusion Criteria:

1. Patients and/or their legal representative must be able to understand the study and voluntarily sign the informed consent form (ICF) per 21 CFR Part 50.55(e)
2. Patients and/or their legal representative accept adherence to protocol requirements
3. Patients who are expected to require parenteral nutrition (PN)for at least 7 days
4. Premature infants (born at 24 to <37 weeks of gestation with a birth weight ≥750g) require at least 80% of targeted energy requirements by PN at study entry (up to 1 month CA); full term infants and children require at least 70% of targeted energy requirements by PN at study entry

Exclusion Criteria:

1. Patients who are not expected to survive hospitalization or with a severe critical unresponsive illness at time of initiation with foreseeable intercurrent events that could jeopardize the patient's participation in the study, as judged by the Investigator (e.g., unresponsive shock, sepsis, renal failure requiring dialysis, severe unresponsive metabolic acidosis, and/or severe unresponsive metabolic disorders);
2. Patients with a known hypersensitivity to lipid emulsion, egg or soybean proteins, or any of the active substances, excipients, or components of the container or who have a history of an adverse event due to ILE;
3. Patients with liver disease including cholestasis;
4. Patients with severe hyperlipidemia or severe disorders of lipid metabolism characterized by hypertriglyceridemia (triglyceride >400 mg/dL);
5. Patients who are unable to tolerate the necessary laboratory monitoring;
6. Patients who are enrolled in another clinical trial involving an investigational agent;
7. Patients with a known history of either severe hemorrhagic or severe hemolytic disease as judged by the investigator;
8. Premature infants born <24 weeks of gestation and patients ≥18 years;
9. Premature infants with a birth weight <750 g;
10. Patient requires or is expected to require propofol for sedation;
11. Patient has received a diagnosis of Coronavirus Disease of 2019 (COVID-19) (diagnosis <2 months prior and/or symptoms have not resolved.
12. Newborn patient born to a mother who was diagnosed as COVID-19 positive at delivery or within 2 months prior to delivery
13. Female patients who are pregnant. Note: All female patients ≥12 years of age must have a negative urine human chorionic gonadotropin (hCG) pregnancy test at screening. For female patients <12 years of age, a urine hCG test at screening will be performed at the discretion of the investigator based on childbearing potential.

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2021-01-22 (Actual); Primary Completion 2022-10-16 (Actual); Study Completion 2022-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Baxter Healthcare Corporation, Study Director — Baxter Healthcare Corporation
Locations (9):
- United States (9):
  - Baxter Investigational Site, Mobile, Alabama
  - Baxter Investigational Site, New Haven, Connecticut
  - Baxter Investigational Site, Orlando, Florida
  - Baxter Investigational Site, Boston, Massachusetts
  - Baxter Investigational Site, Jackson, Mississippi
  - Baxter Investigational Site, Greenville, North Carolina
  - Baxter Investigational Site, Memphis, Tennessee
  - Baxter Investigational Site, San Antonio, Texas
  - Baxter Investigational Site, Provo, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blanco C, Chang W, Bhatt AJ, Gerday E, Talati AJ, Dereddy N, Singh R, Ryan E, Senterre T. Essential fatty acid deficiency, olive oil-based intravenous lipid emulsion, and genetic polymorphisms: A pediatric randomized controlled trial. J Pediatr Gastroenterol Nutr. 2025 Aug;81(2):314-323. doi: 10.1002/jpn3.70072. Epub 2025 May 25. PMID 40415417

RESULTS

PARTICIPANT FLOW:
Groups:
- Clinolipid (Lipid Injectable Emulsion) 20%: Clinolipid was administered intravenously in the hospital setting from 7 up to 90 days using either a syringe pump or an infusion pump as appropriate for the daily volume of infusate. The flow rate was prescribed by the Investigator to provide the daily dosage (based on general pediatric PN guidelines) over 20 to 24 hours and ensure that the maximum lipid infusion rate did not exceed 0.15 g/kg/hour.
- Intralipid (SOC Soybean Oil-based Lipid Emulsion): Intralipid was administered intravenously in the hospital setting from 7 up to 90 days using either a syringe pump or an infusion pump as appropriate for the daily volume of infusate. The flow rate was prescribed by the Investigator to provide the daily dosage (based on general pediatric PN guidelines) over 20 to 24 hours and ensure that the maximum lipid infusion rate did not exceed 0.15 g/kg/hour.
Period: Overall Study
Arm/Group | Clinolipid (Lipid Injectable Emulsion) 20% | Intralipid (SOC Soybean Oil-based Lipid Emulsion)
Started | 50 | 51
Completed | 50 | 50
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population: all patients who were randomized to receive either Clinolipid or standard-of-care soybean oil-based lipid emulsion (Intralipid)
Groups:
- Total: Total of all reporting groups
Arm/Group | Clinolipid (Lipid Injectable Emulsion) 20% | Intralipid (SOC Soybean Oil-based Lipid Emulsion) | Total
Number analyzed (Participants) | 50 | 51 | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 50 | 51 | 101
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Customized [Count of Participants; unit: Participants]
  Pre-Term Neonate (<37 weeks) | 47 | 47 | 94
  Full Term Neonate (=37 weeks to <1 month) | 2 | 2 | 4
  Child (1 to <10 years) | 1 | 1 | 2
  Adolescent (10 to <18 years) | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 29 | 45
  Male | 34 | 22 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 44 | 42 | 86
  Unknown or Not Reported | 3 | 4 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 3
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 21 | 20 | 41
  White | 19 | 23 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 6 | 10
Region of Enrollment [Number; unit: participants]
  United States | 50 | 51 | 101
Weight at birth [Count of Participants; unit: Participants] — Intent-to-treat population: all patients who were randomized to receive either Clinolipid or standard-of-care soybean oil-based lipid emulsion (Intralipid)
  Participants
    Normal (≥ 2500 g) | 1 | 2 | 3
    Low (1500-2499 g) | 4 | 6 | 10
    Very Low (1000-1499 g) | 25 | 28 | 53
    Extremely Low (< 1000 g) | 19 | 13 | 32
    NA ( Child or Adolescent) | 1 | 2 | 3
Diagnosis for PN (NOTE: Multiple diagnoses for PN are allowed, so n may be greater than number of su [Number; unit: participants]
  Prematurity | 46 | 46 | 92
  Gastroschisis | 0 | 3 | 3
  Enteropathies including inflammatory gastrointestinal diseases | 0 | 1 | 1
  Feeding Intolerance | 1 | 0 | 1
  Meconium ileus | 1 | 0 | 1
  Necrotizing enterocolitis | 1 | 0 | 1
  Persistent pulmonary hypertension | 1 | 0 | 1
  Premature infant with feeding intolerance | 1 | 0 | 1
  Premature infant with gastroschisis | 0 | 1 | 2
  Sepsis | 0 | 1 | 1
  Short bowel syndrome | 0 | 1 | 1
  Small for gestational age | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants to Develop Essential Fatty Acid Deficiency (EFAD) Defined by Holman Index > 0.4
Description: Holman Index is the plasma Triene:Tetraene ratio, specifically 5,8,11-eicosatrienoic acid [mead acid] to 5,8,11,14 eicosatetraenoic acid [arachidonic acid, [ARA] ratio
Time Frame: Up to Day 90
Population: Full analysis set: all patients who are randomized to receive either Clinolipid or SoC SO-based lipid emulsion (Intralipid) and have received at least 1 randomized study treatment.
  Per protocol set: all patients in the FAS who have Holman Index measurements taken at baseline and at least 1 other timepoint post-baseline, who have received a minimum of 7 days of ILE treatment, and are without a major protocol violation (i.e., violation that potentially impacts the primary endpoint).
Measure: Count of Participants; unit: Participants
Arm/Group | Clinolipid (Lipid Injectable Emulsion) 20% | Intralipid (SOC Soybean Oil-based Lipid Emulsion)
Number analyzed (Participants) | 50 | 51
Participants | 0 | 0

2. Secondary Outcome: Number of Participants to Develop Parenteral Nutrition-Associated Liver Disease (PNALD)
Description: Defined by direct bilirubin ≥2 mg/dL in patients receiving with intravenous lipid emulsion (ILE).
Time Frame: Up to Day 90
Population: Full analysis set: all patients who are randomized to receive either Clinolipid or SoC SO-based lipid emulsion (Intralipid) and have received at least 1 randomized study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Clinolipid (Lipid Injectable Emulsion) 20% | Intralipid (SOC Soybean Oil-based Lipid Emulsion)
Number analyzed (Participants) | 50 | 51
Participants | 1 | 2

3. Secondary Outcome: Alkaline Phosphatase (ALP)
Description: Plasma liver function test
Time Frame: Up to Day 90
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Clinolipid (Lipid Injectable Emulsion) 20% | Intralipid (SOC Soybean Oil-based Lipid Emulsion)
Number analyzed (Participants) | 50 | 51
IU/L
  Screening: number analyzed (Participants) | 37 | 43
  Screening | 234.0 (98.24) | 187.6 (71.63)
  Baseline (Day 1): number analyzed (Participants) | 12 | 7
  Baseline (Day 1) | 191.9 (62.43) | 239.7 (112.49)
  End of Treatment (EOT): number analyzed (Participants) | 46 | 43
  End of Treatment (EOT) | 405.2 (157.19) | 383.3 (153.87)

4. Secondary Outcome: Aspartate Aminotransferase (AST)
Description: Plasma liver function test
Time Frame: Up to Day 90
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Clinolipid (Lipid Injectable Emulsion) 20% | Intralipid (SOC Soybean Oil-based Lipid Emulsion)
Number analyzed (Participants) | 50 | 51
IU/L
  Screening: number analyzed (Participants) | 37 | 42
  Screening | 44.2 (20.12) | 46.3 (20.76)
  Baseline (Day 1): number analyzed (Participants) | 12 | 7
  Baseline (Day 1) | 45.4 (28.67) | 62.9 (28.00)
  End of Treatment (EOT): number analyzed (Participants) | 46 | 44
  End of Treatment (EOT) | 29.0 (12.40) | 37.7 (28.29)

5. Secondary Outcome: Alanine Aminotransferase (ALT)
Description: Plasma liver function test
Time Frame: Up to Day 90
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Clinolipid (Lipid Injectable Emulsion) 20% | Intralipid (SOC Soybean Oil-based Lipid Emulsion)
Number analyzed (Participants) | 50 | 51
IU/L
  Screening: number analyzed (Participants) | 37 | 42
  Screening | 7.2 (2.79) | 10.3 (9.67)
  Baseline (Day 1): number analyzed (Participants) | 12 | 7
  Baseline (Day 1) | 8.7 (6.88) | 6.7 (0.76)
  End of treatment (EOT): number analyzed (Participants) | 45 | 43
  End of treatment (EOT) | 9.0 (6.48) | 15.3 (26.62)

6. Secondary Outcome: Gamma-Glutamyl Transferase (GGT)
Description: Plasma liver function test
Time Frame: Up to Day 90
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Clinolipid (Lipid Injectable Emulsion) 20% | Intralipid (SOC Soybean Oil-based Lipid Emulsion)
Number analyzed (Participants) | 50 | 51
IU/L
  Screening: number analyzed (Participants) | 33 | 39
  Screening | 97.6 (71.82) | 109.5 (71.14)
  Baseline (Day 1 ): number analyzed (Participants) | 10 | 7
  Baseline (Day 1 ) | 150.1 (76.65) | 120.9 (82.17)
  End of Treatment (EOT): number analyzed (Participants) | 43 | 39
  End of Treatment (EOT) | 109.3 (121.59) | 97.0 (90.39)

7. Secondary Outcome: Total Bilirubin
Description: Plasma liver function test
Time Frame: Up to Day 90
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Clinolipid (Lipid Injectable Emulsion) 20% | Intralipid (SOC Soybean Oil-based Lipid Emulsion)
Number analyzed (Participants) | 50 | 51
umol/L
  Screening: number analyzed (Participants) | 38 | 43
  Screening | 80.065 (36.2491) | 81.133 (51.3912)
  Baseline (Day 1): number analyzed (Participants) | 12 | 7
  Baseline (Day 1) | 78.678 (34.0366) | 80.877 (26.2704)
  End of Treatment (EOT): number analyzed (Participants) | 46 | 44
  End of Treatment (EOT) | 86.944 (44.6590) | 89.948 (50.0126)

8. Secondary Outcome: Direct Bilirubin
Description: Plasma liver function test
Time Frame: Up to Day 90
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Clinolipid (Lipid Injectable Emulsion) 20% | Intralipid (SOC Soybean Oil-based Lipid Emulsion)
Number analyzed (Participants) | 50 | 51
mg/dL
  Screening: number analyzed (Participants) | 34 | 40
  Screening | 0.237 (0.2086) | 0.266 (0.1877)
  Baseline (Day 1): number analyzed (Participants) | 10 | 7
  Baseline (Day 1) | 0.360 (0.0699) | 0.357 (0.0535)
  End of Treatment (EOT): number analyzed (Participants) | 38 | 39
  End of Treatment (EOT) | 0.390 (0.3142) | 0.424 (0.3831)

9. Secondary Outcome: Stigmasterol Blood Level
Description: Phytosterol species
Time Frame: Up to Day 90
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Clinolipid (Lipid Injectable Emulsion) 20% | Intralipid (SOC Soybean Oil-based Lipid Emulsion)
Number analyzed (Participants) | 50 | 51
mg/L
  Baseline (Day 1): number analyzed (Participants) | 43 | 45
  Baseline (Day 1) | 0.80 (1.400) | 1.35 (2.373)
  End of Treatment (EOT): number analyzed (Participants) | 46 | 45
  End of Treatment (EOT) | 0.69 (0.360) | 3.85 (3.077)
  Maximal Value: number analyzed (Participants) | 47 | 44
  Maximal Value | 0.76 (0.542) | 4.07 (3.468)

10. Secondary Outcome: Campesterol Blood Level
Description: Phytosterol species
Time Frame: Up to Day 90
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Clinolipid (Lipid Injectable Emulsion) 20% | Intralipid (SOC Soybean Oil-based Lipid Emulsion)
Number analyzed (Participants) | 50 | 51
mg/dL
  Baseline (Day 1): number analyzed (Participants) | 43 | 45
  Baseline (Day 1) | 1.57 (2.956) | 2.52 (4.510)
  End of Treatment (EOT): number analyzed (Participants) | 46 | 45
  End of Treatment (EOT) | 1.76 (0.787) | 8.11 (6.043)
  Maximal Value: number analyzed (Participants) | 47 | 44
  Maximal Value | 1.89 (1.129) | 8.55 (6.878)

11. Secondary Outcome: Sitosterol Blood Level
Description: Phytosterol species.
Time Frame: Up to day 90
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Clinolipid (Lipid Injectable Emulsion) 20% | Intralipid (SOC Soybean Oil-based Lipid Emulsion)
Number analyzed (Participants) | 50 | 51
mg/L
  Baseline (Day 1): number analyzed (Participants) | 43 | 45
  Baseline (Day 1) | 4.51 (8.223) | 8.06 (15.782)
  End of Treatment (EOT): number analyzed (Participants) | 46 | 44
  End of Treatment (EOT) | 17.89 (9.499) | 23.40 (17.560)
  Maximal Value: number analyzed (Participants) | 47 | 44
  Maximal Value | 20.09 (17.225) | 26.05 (22.180)

12. Secondary Outcome: Cholesterol Blood Level
Time Frame: Up to Day 90
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Clinolipid (Lipid Injectable Emulsion) 20% | Intralipid (SOC Soybean Oil-based Lipid Emulsion)
Number analyzed (Participants) | 50 | 51
mmol/L
  Baseline (Day 1): number analyzed (Participants) | 43 | 46
  Baseline (Day 1) | 2.521 (0.7933) | 2.537 (0.9566)
  End of Treatment (EOT): number analyzed (Participants) | 45 | 47
  End of Treatment (EOT) | 3.019 (0.6337) | 2.773 (0.6801)
  Maximal Value: number analyzed (Participants) | 45 | 47
  Maximal Value | 3.194 (1.2764) | 2.799 (0.6884)

13. Secondary Outcome: Squalene Blood Level
Time Frame: Up to Day 90
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Clinolipid (Lipid Injectable Emulsion) 20% | Intralipid (SOC Soybean Oil-based Lipid Emulsion)
Number analyzed (Participants) | 50 | 51
mg/L
  Baseline (Day 1): number analyzed (Participants) | 43 | 45
  Baseline (Day 1) | 0.28 (0.735) | 0.13 (0.130)
  End of Treatment (EOT): number analyzed (Participants) | 46 | 45
  End of Treatment (EOT) | 0.50 (0.778) | 0.30 (0.213)
  Maximal Value: number analyzed (Participants) | 47 | 44
  Maximal Value | 0.54 (0.777) | 0.30 (0.213)

14. Secondary Outcome: Calories Nutritional Intake
Time Frame: Up to Day 90
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kCal/kg/24 hours
Arm/Group | Clinolipid (Lipid Injectable Emulsion) 20% | Intralipid (SOC Soybean Oil-based Lipid Emulsion)
Number analyzed (Participants) | 50 | 51
kCal/kg/24 hours
  Parenteral Nutrition(PN), Screening: number analyzed (Participants) | 35 | 36
  Parenteral Nutrition(PN), Screening | 45.1 (17.19) | 44.1 (18.41)
  PN, Baseline (Day 1) | 42.3 (22.29) | 45.4 (24.42)
  PN, Day 2 | 57 (15.71) | 57.4 (17.18)
  PN, Day 3: number analyzed (Participants) | 49 | 49
  PN, Day 3 | 59.1 (14.47) | 63.1 (17.17)
  PN, Day 4: number analyzed (Participants) | 49 | 47
  PN, Day 4 | 58.0 (15.76) | 62.2 (16.73)
  PN, Day 5: number analyzed (Participants) | 49 | 47
  PN, Day 5 | 54.7 (19.09) | 55.4 (19.60)
  PN, Day 6: number analyzed (Participants) | 46 | 46
  PN, Day 6 | 48.6 (20.45) | 50.8 (20.44)
  PN, Day 7: number analyzed (Participants) | 41 | 39
  PN, Day 7 | 45.5 (24.84) | 47.6 (24.42)
  PN, Day 8: number analyzed (Participants) | 17 | 18
  PN, Day 8 | 58.0 (28.60) | 60.40 (24.51)
  PN, Day 9: number analyzed (Participants) | 15 | 15
  PN, Day 9 | 59.3 (27.28) | 62.2 (25.60)
  PN, Day 10: number analyzed (Participants) | 10 | 14
  PN, Day 10 | 64.4 (22.94) | 60.7 (30.08)
  PN, Day 11: number analyzed (Participants) | 9 | 12
  PN, Day 11 | 61.6 (17.08) | 61.2 (25.49)
  PN, Day 12: number analyzed (Participants) | 9 | 11
  PN, Day 12 | 53.0 (17.87) | 60.8 (28.16)
  PN, Day 13: number analyzed (Participants) | 8 | 11
  PN, Day 13 | 48.4 (22.24) | 53.4 (31.88)
  PN, Day 14: number analyzed (Participants) | 4 | 9
  PN, Day 14 | 62.4 (34.32) | 63.4 (27.85)
  PN, Day 90/EOT: number analyzed (Participants) | 10 | 11
  PN, Day 90/EOT | 34.3 (15.53) | 42.6 (23.76)
  Enteral Nutrition (EN), Screening: number analyzed (Participants) | 13 | 11
  Enteral Nutrition (EN), Screening | 14.2 (14.00) | 8.0 (5.29)
  EN, Baseline Day 1: number analyzed (Participants) | 33 | 32
  EN, Baseline Day 1 | 10.6 (7.82) | 8.8 (6.25)
  EN, Day 2: number analyzed (Participants) | 45 | 40
  EN, Day 2 | 15.4 (10.57) | 14.6 (7.74)
  EN, Day 3: number analyzed (Participants) | 44 | 38
  EN, Day 3 | 19.8 (11.99) | 19.6 (12.54)
  EN, Day 4: number analyzed (Participants) | 42 | 39
  EN, Day 4 | 29.2 (16.78) | 23.8 (15.96)
  EN, Day 5: number analyzed (Participants) | 43 | 39
  EN, Day 5 | 38.9 (18.50) | 34.3 (18.14)
  EN, Day 6: number analyzed (Participants) | 42 | 39
  EN, Day 6 | 42.9 (24.24) | 43.2 (21.34)
  EN, Day 7: number analyzed (Participants) | 37 | 36
  EN, Day 7 | 50.8 (28.40) | 52.3 (25.06)
  EN, Day 8: number analyzed (Participants) | 15 | 12
  EN, Day 8 | 35.5 (25.63) | 36.4 (25.84)
  EN, Day 9: number analyzed (Participants) | 13 | 8
  EN, Day 9 | 37.6 (24.47) | 40.9 (22.83)
  EN, Day 10: number analyzed (Participants) | 10 | 7
  EN, Day 10 | 32.0 (26.29) | 52.2 (24.35)
  EN, Day 11: number analyzed (Participants) | 8 | 8
  EN, Day 11 | 34.4 (14.73) | 34.3 (27.46)
  EN, Day 12: number analyzed (Participants) | 8 | 8
  EN, Day 12 | 47.2 (14.67) | 34.6 (24.06)
  EN, Day 13: number analyzed (Participants) | 7 | 9
  EN, Day 13 | 50.3 (24.12) | 33.5 (23.24)
  EN, Day 14: number analyzed (Participants) | 4 | 7
  EN, Day 14 | 30.8 (36.74) | 35.6 (26.30)
  EN, Day 90/EOT: number analyzed (Participants) | 38 | 36
  EN, Day 90/EOT | 84.4 (17.92) | 73.3 (24.56)
  Intravenous (IV) Fluids, Screening: number analyzed (Participants) | 18 | 20
  Intravenous (IV) Fluids, Screening | 20.0 (10.60) | 22.0 (10.02)
  IV Fluids, Baseline (Day 1): number analyzed (Participants) | 5 | 4
  IV Fluids, Baseline (Day 1) | 18.3 (12.74) | 21.0 (13.21)
  IV, Fluids, Day 2: number analyzed (Participants) | 2 | 1
  IV, Fluids, Day 2 | 16.7 (12.34) | 33.1 (NA) — Standard Deviation is not calculable for 1 participant
  IV, Fluids, Day 3: number analyzed (Participants) | 0 | 1
  IV, Fluids, Day 3 |  | 0.5 (NA) — Standard Deviation is not calculable for 1 participant
  IV, Fluids, Day 5: number analyzed (Participants) | 0 | 1
  IV, Fluids, Day 5 |  | 30.2 (NA) — Standard Deviation is not calculable for 1 participant
  IV, Fluids, Day 6: number analyzed (Participants) | 1 | 0
  IV, Fluids, Day 6 | 8.9 (NA) — Standard Deviation is not calculable for 1 participant |
  IV, Fluids, Day 7: number analyzed (Participants) | 0 | 1
  IV, Fluids, Day 7 |  | 9.3 (NA) — Standard Deviation is not calculable for 1 participant
  IV, Fluids, Day 90:EOT: number analyzed (Participants) | 2 | 0
  IV, Fluids, Day 90:EOT | 5.6 (3.92) |

15. Secondary Outcome: Protein Nutritional Intake
Time Frame: Up to Day 90
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g/kg/24hours
Arm/Group | Clinolipid (Lipid Injectable Emulsion) 20% | Intralipid (SOC Soybean Oil-based Lipid Emulsion)
Number analyzed (Participants) | 50 | 51
g/kg/24hours
  Parenteral (PN), Screening: number analyzed (Participants) | 34 | 35
  Parenteral (PN), Screening | 3.33 (2.375) | 3.20 (2.024)
  PN, Baseline (Day 1) | 2.45 (1.106) | 2.56 (1.116)
  PN, Day 2 | 2.78 (0.732) | 2.83 (0.711)
  PN, Day 3: number analyzed (Participants) | 49 | 49
  PN, Day 3 | 2.74 (0.737) | 2.86 (0.694)
  PN, Day 4: number analyzed (Participants) | 49 | 47
  PN, Day 4 | 2.61 (0.709) | 2.81 (0.646)
  PN, Day 5: number analyzed (Participants) | 49 | 47
  PN, Day 5 | 2.43 (0.858) | 2.53 (0.801)
  PN, Day 6: number analyzed (Participants) | 46 | 46
  PN, Day 6 | 2.25 (0.905) | 2.35 (0.880)
  PN, Day 7: number analyzed (Participants) | 41 | 39
  PN, Day 7 | 2.08 (1.046) | 2.18 (1.039)
  PN, Day 8: number analyzed (Participants) | 17 | 18
  PN, Day 8 | 2.57 (1.141) | 2.83 (1.007)
  PN, Day 9: number analyzed (Participants) | 15 | 15
  PN, Day 9 | 2.57 (1.080) | 2.97 (1.121)
  PN, Day 10: number analyzed (Participants) | 11 | 14
  PN, Day 10 | 2.71 (0.888) | 2.88 (1.064)
  PN, Day 11: number analyzed (Participants) | 9 | 12
  PN, Day 11 | 2.53 (0.902) | 2.78 (0.880)
  PN, Day 12: number analyzed (Participants) | 9 | 11
  PN, Day 12 | 2.31 (1.039) | 2.75 (0.969)
  PN, Day 13: number analyzed (Participants) | 8 | 11
  PN, Day 13 | 2.16 (1.163) | 2.43 (1.240)
  PN, Day 14: number analyzed (Participants) | 4 | 9
  PN, Day 14 | 2.37 (1.315) | 2.76 (0.969)
  PN, Day 90 EOT: number analyzed (Participants) | 10 | 11
  PN, Day 90 EOT | 2.02 (1.245) | 1.98 (0.596)
  Enteral Nutrition (EN), Screening: number analyzed (Participants) | 13 | 11
  Enteral Nutrition (EN), Screening | 0.33 (0.480) | 0.14 (0.087)
  EN, Baseline ( Day 1): number analyzed (Participants) | 33 | 32
  EN, Baseline ( Day 1) | 0.22 (0.209) | 0.15 (0.106)
  EN, Day 2: number analyzed (Participants) | 45 | 40
  EN, Day 2 | 0.34 (0.389) | 0.26 (0.136)
  EN, Day 3: number analyzed (Participants) | 44 | 38
  EN, Day 3 | 0.42 (0.395) | 0.35 (0.223)
  EN, Day 4: number analyzed (Participants) | 42 | 39
  EN, Day 4 | 0.59 (0.499) | 0.44 (0.328)
  EN, Day 5: number analyzed (Participants) | 43 | 39
  EN, Day 5 | 0.79 (0.548) | 0.63 (0.358)
  EN, Day 6: number analyzed (Participants) | 43 | 39
  EN, Day 6 | 0.89 (0.599) | 0.80 (0.423)
  EN, Day 7: number analyzed (Participants) | 37 | 36
  EN, Day 7 | 1.04 (0.668) | 0.95 (0.461)
  EN, Day 8: number analyzed (Participants) | 15 | 12
  EN, Day 8 | 0.68 (0.478) | 0.66 (0.454)
  EN, Day 9: number analyzed (Participants) | 13 | 8
  EN, Day 9 | 0.69 (0.430) | 0.81 (0.435)
  EN, Day 10: number analyzed (Participants) | 10 | 7
  EN, Day 10 | 0.56 (0.430) | 0.93 (0.466)
  EN, Day 11: number analyzed (Participants) | 8 | 8
  EN, Day 11 | 0.68 (0.304) | 0.59 (0.442)
  EN, Day 12: number analyzed (Participants) | 8 | 8
  EN, Day 12 | 0.96 (0.475) | 0.59 (0.404)
  EN, Day 13: number analyzed (Participants) | 7 | 9
  EN, Day 13 | 1.04 (0.731) | 0.67 (0.490)
  EN, Day 14: number analyzed (Participants) | 3 | 7
  EN, Day 14 | 0.76 (0.795) | 0.54 (0.309)
  EN, Day 90/EOT: number analyzed (Participants) | 37 | 37
  EN, Day 90/EOT | 1.69 (0.659) | 1.34 (0.427)

16. Secondary Outcome: Lipid Nutritional Intake
Time Frame: Up to Day 90
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g/kg/24 hours
Arm/Group | Clinolipid (Lipid Injectable Emulsion) 20% | Intralipid (SOC Soybean Oil-based Lipid Emulsion)
Number analyzed (Participants) | 50 | 51
g/kg/24 hours
  Parenteral Nutrition (PN), Screening: number analyzed (Participants) | 21 | 23
  Parenteral Nutrition (PN), Screening | 1.56 (0.584) | 1.84 (0.691)
  PN, Baseline (Day 1) | 1.74 (0.855) | 1.76 (0.944)
  PN, Day 2 | 2.48 (0.692) | 2.55 (0.751)
  PN, Day 3: number analyzed (Participants) | 47 | 49
  PN, Day 3 | 3.07 (0.713) | 3.14 (0.592)
  PN, Day 4: number analyzed (Participants) | 49 | 47
  PN, Day 4 | 2.96 (0.690) | 3.17 (0.520)
  PN, Day 5: number analyzed (Participants) | 49 | 47
  PN, Day 5 | 2.78 (0.673) | 2.81 (0.628)
  PN, Day 6: number analyzed (Participants) | 46 | 46
  PN, Day 6 | 2.38 (0.857) | 2.33 (0.927)
  PN, Day 7: number analyzed (Participants) | 41 | 42
  PN, Day 7 | 2.15 (1.026) | 2.22 (1.032)
  PN, Day 8: number analyzed (Participants) | 17 | 18
  PN, Day 8 | 2.92 (0.598) | 2.91 (0.746)
  PN, Day 9: number analyzed (Participants) | 15 | 15
  PN, Day 9 | 2.64 (0.751) | 2.97 (0.520)
  PN, Day 10: number analyzed (Participants) | 11 | 14
  PN, Day 10 | 2.73 (0.763) | 3.00 (0.735)
  PN, Day 11: number analyzed (Participants) | 9 | 12
  PN, Day 11 | 2.97 (0.494) | 3.07 (0.884)
  PN, Day 12: number analyzed (Participants) | 9 | 11
  PN, Day 12 | 2.78 (0.592) | 3.13 (0.497)
  PN, Day 13: number analyzed (Participants) | 8 | 11
  PN, Day 13 | 2.70 (0.678) | 2.82 (0.973)
  PN, Day 14: number analyzed (Participants) | 4 | 9
  PN, Day 14 | 3.30 (0.480) | 2.78 (0.829)
  PN, Day 90/ EOT: number analyzed (Participants) | 3 | 4
  PN, Day 90/ EOT | 1.50 (0.863) | 2.27 (1.290)
  Enteral Nutrition (EN), Screening: number analyzed (Participants) | 13 | 11
  Enteral Nutrition (EN), Screening | 0.71 (0.614) | 0.42 (0.260)
  EN, Baseline (Day 1): number analyzed (Participants) | 33 | 32
  EN, Baseline (Day 1) | 0.58 (0.459) | 0.46 (0.319)
  EN, Day 2: number analyzed (Participants) | 45 | 40
  EN, Day 2 | 0.88 (0.741) | 0.77 (0.409)
  EN, Day 3: number analyzed (Participants) | 44 | 38
  EN, Day 3 | 1.14 (0.844) | 1.04 (0.688)
  EN, Day 4: number analyzed (Participants) | 42 | 39
  EN, Day 4 | 1.62 (1.073) | 1.27 (0.828)
  EN, Day 5: number analyzed (Participants) | 43 | 39
  EN, Day 5 | 2.18 (1.168) | 1.81 (0.935)
  EN, Day 6: number analyzed (Participants) | 43 | 39
  EN, Day 6 | 2.30 (1.279) | 2.21 (0.990)
  EN, Day 7: number analyzed (Participants) | 37 | 36
  EN, Day 7 | 2.68 (1.436) | 2.66 (1.164)
  EN, Day 8: number analyzed (Participants) | 15 | 12
  EN, Day 8 | 1.79 (1.190) | 1.88 (1.185)
  EN, Day 9: number analyzed (Participants) | 13 | 8
  EN, Day 9 | 1.85 (1.142) | 2.17 (1.035)
  EN, Day 10: number analyzed (Participants) | 10 | 7
  EN, Day 10 | 1.59 (1.213) | 2.49 (1.026)
  EN, Day 11: number analyzed (Participants) | 8 | 8
  EN, Day 11 | 1.82 (0.802) | 1.73 (1.274)
  EN, Day 12: number analyzed (Participants) | 8 | 8
  EN, Day 12 | 2.46 (0.833) | 1.74 (1.184)
  EN, Day 13: number analyzed (Participants) | 7 | 9
  EN, Day 13 | 2.51 (1.149) | 1.89 (1.300)
  EN, Day 14: number analyzed (Participants) | 3 | 7
  EN, Day 14 | 1.92 (1.809) | 1.61 (0.882)
  EN, Day 90 EOT: number analyzed (Participants) | 37 | 36
  EN, Day 90 EOT | 4.33 (1.058) | 3.71 (1.070)

17. Secondary Outcome: Carbohydrates Nutritional Intake
Time Frame: Up to Day 90
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g/kg/24 hours
Arm/Group | Clinolipid (Lipid Injectable Emulsion) 20% | Intralipid (SOC Soybean Oil-based Lipid Emulsion)
Number analyzed (Participants) | 50 | 51
g/kg/24 hours
  Parenteral Nutrition (PN) Screening: number analyzed (Participants) | 35 | 36
  Parenteral Nutrition (PN) Screening | 7.61 (2.248) | 7.47 (3.087)
  PN, Baseline (Day 1) | 6.41 (3.309) | 6.99 (3.710)
  PN, Day 2 | 8.52 (2.524) | 8.51 (2.894)
  PN, Day 3: number analyzed (Participants) | 49 | 49
  PN, Day 3 | 8.78 (2.457) | 9.05 (2.950)
  PN, Day 4: number analyzed (Participants) | 49 | 47
  PN, Day 4 | 8.50 (2.695) | 9.13 (3.025)
  PN, Day 5: number analyzed (Participants) | 49 | 47
  PN, Day 5 | 8.24 (3.083) | 8.51 (3.216)
  PN, Day 6: number analyzed (Participants) | 46 | 46
  PN, Day 6 | 7.47 (3.397) | 8.19 (3.265)
  PN, Day 7: number analyzed (Participants) | 41 | 39
  PN, Day 7 | 7.30 (3.850) | 7.77 (3.746)
  PN, Day 8: number analyzed (Participants) | 17 | 18
  PN, Day 8 | 9.15 (4.479) | 8.96 (4.260)
  PN, Day 9: number analyzed (Participants) | 15 | 15
  PN, Day 9 | 9.40 (4.144) | 9.00 (4.700)
  PN, Day 10: number analyzed (Participants) | 11 | 14
  PN, Day 10 | 9.99 (3.451) | 9.21 (4.840)
  PN, Day 11: number analyzed (Participants) | 9 | 12
  PN, Day 11 | 8.79 (2.723) | 9.47 (4.123)
  PN, Day 12: number analyzed (Participants) | 9 | 11
  PN, Day 12 | 7.45 (2.337) | 9.47 (4.697)
  PN, Day 13: number analyzed (Participants) | 8 | 11
  PN, Day 13 | 6.65 (3.077) | 8.58 (5.046)
  PN, Day 14: number analyzed (Participants) | 4 | 9
  PN, Day 14 | 10.30 (5.276) | 10.20 (4.836)
  PN, Day 90/EOT: number analyzed (Participants) | 10 | 11
  PN, Day 90/EOT | 6.34 (2.535) | 8.10 (3.815)
  Enteral Nutrition (EN), Screening: number analyzed (Participants) | 13 | 11
  Enteral Nutrition (EN), Screening | 1.58 (1.657) | 0.86 (0.534)
  EN, Baseline (Day 1): number analyzed (Participants) | 33 | 32
  EN, Baseline (Day 1) | 1.19 (0.893) | 0.95 (0.656)
  EN, Day 2: number analyzed (Participants) | 45 | 40
  EN, Day 2 | 1.70 (1.195) | 1.59 (0.841)
  EN, Day 3: number analyzed (Participants) | 44 | 38
  EN, Day 3 | 2.21 (1.362) | 2.14 (1.372)
  EN, Day 4: number analyzed (Participants) | 42 | 39
  EN, Day 4 | 3.14 (1.765) | 2.64 (1.757)
  EN, Day 5: number analyzed (Participants) | 43 | 39
  EN, Day 5 | 4.28 (1.968) | 3.75 (1.971)
  EN, Day 6: number analyzed (Participants) | 43 | 39
  EN, Day 6 | 4.64 (2.413) | 4.63 (2.123)
  EN, Day 7: number analyzed (Participants) | 37 | 36
  EN, Day 7 | 5.40 (2.731) | 5.54 (2.463)
  EN, Day 8: number analyzed (Participants) | 15 | 12
  EN, Day 8 | 3.80 (2.519) | 3.89 (2.500)
  EN, Day 9: number analyzed (Participants) | 13 | 8
  EN, Day 9 | 3.92 (2.377) | 4.56 (2.217)
  EN, Day 10: number analyzed (Participants) | 10 | 7
  EN, Day 10 | 3.31 (2.514) | 5.23 (2.247)
  EN, Day 11: number analyzed (Participants) | 8 | 8
  EN, Day 11 | 3.87 (1.615) | 3.56 (2.635)
  EN, Day 12: number analyzed (Participants) | 8 | 8
  EN, Day 12 | 5.29 (1.851) | 3.59 (2.443)
  EN, Day 13: number analyzed (Participants) | 7 | 9
  EN, Day 13 | 5.51 (2.766) | 3.94 (2.733)
  EN, Day 14: number analyzed (Participants) | 3 | 7
  EN, Day 14 | 4.10 (3.944) | 3.31 (1.827)
  EN, Day 90/EOT: number analyzed (Participants) | 37 | 36
  EN, Day 90/EOT | 8.77 (1.695) | 7.75 (2.249)
  Intravenous (IV) Fluids, Screening: number analyzed (Participants) | 18 | 20
  Intravenous (IV) Fluids, Screening | 5.88 (3.119) | 6.47 (2.947)
  IV Fluids, Baseline (Day 1): number analyzed (Participants) | 5 | 4
  IV Fluids, Baseline (Day 1) | 5.37 (3.748) | 6.19 (3.886)
  IV Fluids, Day 2: number analyzed (Participants) | 2 | 1
  IV Fluids, Day 2 | 4.92 (3.628) | 9.74 (NA) — Standard Deviation is not calculable for 1 participant
  IV Fluids, Day 3: number analyzed (Participants) | 0 | 1
  IV Fluids, Day 3 |  | 0.14 (NA) — Standard Deviation is not calculable for 1 participant
  IV Fluids, Day 5: number analyzed (Participants) | 0 | 1
  IV Fluids, Day 5 |  | 8.89 (NA) — Standard Deviation is not calculable for 1 participant
  IV Fluids, Day 6: number analyzed (Participants) | 1 | 0
  IV Fluids, Day 6 | 2.62 (NA) — Standard Deviation is not calculable for 1 participant |
  IV Fluids, Day 7: number analyzed (Participants) | 0 | 1
  IV Fluids, Day 7 |  | 2.72 (NA) — Standard Deviation is not calculable for 1 participant
  IV Fluids, Day 90/EOT: number analyzed (Participants) | 2 | 0
  IV Fluids, Day 90/EOT | 1.63 (1.153) |

18. Secondary Outcome: Change in Length or Height (and Head Circumference for Infants <1 Year of Age) From Baseline
Description: Change in length/height from baseline (mm/week in all) = [Length (mm) on Day X - Length (mm) at baseline] / [X/7] Change in head circumference from baseline (mm/week in infants <1 year) = [Head circumference (mm) on Day X - Head circumference (mm) at baseline] / [X/7]
Time Frame: Up to Day 90
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm/week
Arm/Group | Clinolipid (Lipid Injectable Emulsion) 20% | Intralipid (SOC Soybean Oil-based Lipid Emulsion)
Number analyzed (Participants) | 50 | 51
mm/week
  Change in Length or Height from Baseline to Day 90/EOT: number analyzed (Participants) | 48 | 45
  Change in Length or Height from Baseline to Day 90/EOT | 13.298 (15.4004) | 6.406 (8.6426)
  Change in Head Circumference from Baseline to Day 90/EOT for Infants < 1 Year of Age: number analyzed (Participants) | 49 | 45
  Change in Head Circumference from Baseline to Day 90/EOT for Infants < 1 Year of Age | 0.918 (6.5248) | -0.218 (5.6635)

19. Secondary Outcome: Body Weight
Description: Change in Weight. from baseline (g/kg/day) to EOT for infants < 1 year of Age
Time Frame: Up to day 90
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g/kg/day
Arm/Group | Clinolipid (Lipid Injectable Emulsion) 20% | Intralipid (SOC Soybean Oil-based Lipid Emulsion)
Number analyzed (Participants) | 46 | 44
g/kg/day | 7.372 (10.1814) | 5.435 (11.8946)

20. Secondary Outcome: Body Weight
Description: Change in weight from baseline to end of treatment (EOT) for those > 1 year of age (g/day)
Time Frame: Upto Day 90
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g/day
Arm/Group | Clinolipid (Lipid Injectable Emulsion) 20% | Intralipid (SOC Soybean Oil-based Lipid Emulsion)
Number analyzed (Participants) | 1 | 2
g/day | 71.429 (NA) — Standard Deviation is not calculable for 1 participant | -100.000 (141.4214)

21. Secondary Outcome: Number of Adverse Events of Special Interest
Time Frame: Up to Day 120 (30 Days After Subject's Last Study Treatment if hospital discharge has not occurred)
Population: Safety analysis set (SS): the set of all patients who have been administered study treatment (Clinolipid or Intralipid). Patients will be analyzed according to treatment received.
Measure: Number; unit: Number of Events per 100 Patient Days
Arm/Group | Clinolipid (Lipid Injectable Emulsion) 20% | Intralipid (SOC Soybean Oil-based Lipid Emulsion)
Number analyzed (Participants) | 50 | 51
Number of Events per 100 Patient Days
  COAGULATION FACTOR DEFICIENCY | 0 | 0.2
  VOMITING | 0.4 | 0
  CATHETER SITE ULCER | 0 | 0.2
  INFUSION SITE EXTRAVASATION | 0 | 0.2
  ACUTE RESPIRATORY FAILURE | 0.2 | 0
  BRONCHOPULMONARY DYSPLASIA | 0.4 | 0.2
  DYSPNOEA | 0.2 | 0
  HYPOXIA | 0 | 0.2
  INFANTILE APNOEA | 0.6 | 0.7
  NEONATAL RESPIRATORY DISTRESS | 0 | 0.2
  STRIDOR | 0.2 | 0

22. Secondary Outcome: Number of Participants With Neonatal Morbidities
Description: Neonatal Morbidities are presented for premature infants born < 37 weeks of gestation up to 1 month corrected age. Patients may have more than 1 neonatal morbidity.
Time Frame: Up to Day 90
Measure: Count of Participants; unit: Participants
Arm/Group | Clinolipid (Lipid Injectable Emulsion) 20% | Intralipid (SOC Soybean Oil-based Lipid Emulsion)
Number analyzed (Participants) | 50 | 51
Participants
  Any Neonatal Morbidity | 13 | 7
  Bronchopulmonary dysplasia | 2 | 1
  Retinopathy of prematurity | 1 | 0
  Intraventricular hemorrhage | 7 | 6
  Necrotizing enterocolitis | 1 | 0
  Late-onset sepsis | 2 | 0

ADVERSE EVENTS:
Time Frame: Up to day 120
Arm/Group | Clinolipid (Lipid Injectable Emulsion) 20% | Intralipid (SOC Soybean Oil-based Lipid Emulsion)
All-Cause Mortality (participants affected / at risk) | 1/50 | 0/51
Serious Adverse Events (participants affected / at risk) | 2/50 | 2/51
Other Adverse Events (participants affected / at risk) | 40/50 | 39/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clinolipid (Lipid Injectable Emulsion) 20% (N=50) | Intralipid (SOC Soybean Oil-based Lipid Emulsion) (N=51)
PNEUMOPERITONEUM (Gastrointestinal disorders) | 0 | 1
HYPOXIC-ISCHAEMIC ENCEPHALOPATHY (Nervous system disorders) | 1 | 0
INTRAVENTRICULAR HAEMORRHAGE NEONATAL (Nervous system disorders) | 0 | 1
SEIZURE (Nervous system disorders) | 0 | 1
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clinolipid (Lipid Injectable Emulsion) 20% (N=50) | Intralipid (SOC Soybean Oil-based Lipid Emulsion) (N=51)
ANAEMIA NEONATAL (Blood and lymphatic system disorders) | 14 | 15
COAGULATION FACTOR DEFICIENCY (Blood and lymphatic system disorders) | 0 | 1
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 | 1
BRADYCARDIA NEONATAL (Cardiac disorders) | 3 | 2
CARDIAC DYSFUNCTION (Cardiac disorders) | 0 | 1
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 | 0
ADRENAL INSUFFICIENCY NEONATAL (Congenital, familial and genetic disorders) | 2 | 2
ANKYLOGLOSSIA CONGENITAL (Congenital, familial and genetic disorders) | 0 | 1
ATRIAL SEPTAL DEFECT (Congenital, familial and genetic disorders) | 5 | 5
HYDROCELE (Congenital, familial and genetic disorders) | 2 | 0
NEWBORN PERSISTENT PULMONARY HYPERTENSION (Congenital, familial and genetic disorders) | 1 | 1
PATENT DUCTUS ARTERIOSUS (Congenital, familial and genetic disorders) | 15 | 8
PHYTOSTEROLAEMIA (Congenital, familial and genetic disorders) | 0 | 1
PSEUDOHYPOALDOSTERONISM (Congenital, familial and genetic disorders) | 0 | 1
HYPOTHYROIDISM (Endocrine disorders) | 1 | 0
EYE DISCHARGE (Eye disorders) | 1 | 1
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 | 3
ANAL FISSURE (Gastrointestinal disorders) | 1 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2 | 1
HAEMATOCHEZIA (Gastrointestinal disorders) | 2 | 0
Ileus (Gastrointestinal disorders) | 0 | 2
INTESTINAL DILATATION (Gastrointestinal disorders) | 0 | 1
MECONIUM PLUG SYNDROME (Gastrointestinal disorders) | 1 | 0
NECROTISING ENTEROCOLITIS NEONATAL (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
ADMINISTRATION SITE EXTRAVASATION (General disorders) | 1 | 0
CATHETER SITE ULCER (General disorders) | 0 | 1
INFUSION SITE EXTRAVASATION (General disorders) | 1 | 4
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 | 3
HYPERBILIRUBINAEMIA NEONATAL (Hepatobiliary disorders) | 22 | 20
CONJUNCTIVITIS (Infections and infestations) | 0 | 1
EYE INFECTION (Infections and infestations) | 1 | 0
PUSTULE (Infections and infestations) | 0 | 1
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 0 | 1
SEPSIS NEONATAL (Infections and infestations) | 5 | 2
SKIN INFECTION (Infections and infestations) | 0 | 1
STREPTOCOCCAL SEPSIS (Infections and infestations) | 0 | 1
TRACHEITIS (Infections and infestations) | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 3 | 2
URINARY TRACT INFECTION FUNGAL (Infections and infestations) | 1 | 0
URINARY TRACT INFECTION NEONATAL (Infections and infestations) | 1 | 0
WOUND INFECTION (Infections and infestations) | 0 | 2
POSTOPERATIVE RESPIRATORY FAILURE (Injury, poisoning and procedural complications) | 1 | 0
SKIN ABRASION (Injury, poisoning and procedural complications) | 0 | 2
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 5 | 3
BLOOD TRIGLYCERIDES INCREASED (Investigations) | 2 | 0
CARDIOVASCULAR EXAMINATION ABNORMAL (Investigations) | 1 | 0
FREE FATTY ACIDS DECREASED (Investigations) | 1 | 0
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 | 2
GASTRIC FLUID ANALYSIS ABNORMAL (Investigations) | 1 | 0
PHYTOSTEROL LEVEL INCREASED (Investigations) | 1 | 0
TRANSAMINASES INCREASED (Investigations) | 0 | 1
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 0 | 1
FEEDING INTOLERANCE (Metabolism and nutrition disorders) | 7 | 3
HYPERCHLORAEMIA (Metabolism and nutrition disorders) | 2 | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 1
HYPERMAGNESAEMIA (Metabolism and nutrition disorders) | 1 | 1
HYPERNATRAEMIA (Metabolism and nutrition disorders) | 2 | 3
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 1 | 2
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 0 | 2
NEONATAL HYPONATRAEMIA (Metabolism and nutrition disorders) | 5 | 7
OSTEOPENIA (Musculoskeletal and connective tissue disorders) | 2 | 2
HAEMANGIOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
HYDROCEPHALUS (Nervous system disorders) | 1 | 0
INTRAVENTRICULAR HAEMORRHAGE (Nervous system disorders) | 0 | 2
INTRAVENTRICULAR HAEMORRHAGE NEONATAL (Nervous system disorders) | 6 | 5
RENAL INJURY (Renal and urinary disorders) | 1 | 0
BRONCHOPULMONARY DYSPLASIA (Respiratory, thoracic and mediastinal disorders) | 2 | 3
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
INFANTILE APNOEA (Respiratory, thoracic and mediastinal disorders) | 5 | 3
NEONATAL RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
NEONATAL RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 | 0
STRIDOR (Respiratory, thoracic and mediastinal disorders) | 1 | 0
DERMATITIS DIAPER (Skin and subcutaneous tissue disorders) | 2 | 2
RASH (Skin and subcutaneous tissue disorders) | 0 | 1
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 1 | 0
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 0 | 1
SKIN DISORDER (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor reserves the right of prior review and approval of data from this study relative to the potential release of proprietary information to any publication or for any presentation.

DOCUMENTS (2):
  • Study Protocol (2022-02-22): https://cdn.clinicaltrials.gov/large-docs/44/NCT04555044/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-30): https://cdn.clinicaltrials.gov/large-docs/44/NCT04555044/SAP_001.pdf